CLINICAL TRIAL: NCT05530486
Title: Effect of the Use of Therapeutic Low-intensity 660 nm LASER in the Treatment of Diabetic Ulcers: a Double-blind Randomized Clinical Trial
Brief Title: Effect of the Use of Low Intensity Therapeutic LASER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Piaui (Other)
Responsible Party: Principal Investigator, Vinicius Saura Cardoso, principal investigator, Federal University of Piaui
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 5.588.474
Record Dates: First submitted 2022-09-01; First posted 2022-09-07 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-03

CONDITIONS: Wound; Diabetic Foot; LTBI
Keywords: Diabetes Mellitus; Low-Level Light Therapy; Diabetic Foot
MeSH Terms: conditions — Wounds and Injuries; Diabetic Foot; Diabetes Mellitus | interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Comparador de placebo: CC + curativo (Placebo Comparator): The group will receive placebo LASER application associated with Helianthus annuus oil dressing.
  Interventions: Device: CC; Procedure: Dressing
- Comparador ativo: LG1 + curativo (Active Comparator): The group will receive application of LASER Gallium Arsenide (GasAs) 660 nm 4 J/cm² associated with Helianthus annuus oil dressing.
  Interventions: Device: LG1; Procedure: Dressing
- Comparador ativo: LG2 + curativo (Active Comparator): The group will receive application of LASER Gallium Arsenide (GaAs) 660 nm 8 J/cm² associated with Helianthus annuus oil dressing.
  Interventions: Device: LG2; Procedure: Dressing
- Comparador ativo: LG3 + curativo (Active Comparator): The group will receive application of LASER Gallium Arsenide (GaAs) 660 nm 12 J/cm² associated with Helianthus annuus oil dressing.
  Interventions: Device: LG3; Procedure: Dressing

INTERVENTIONS:
Device: CC — Application of placebo LASER
  Arms: Comparador de placebo: CC + curativo
Device: LG1 — Application of LASER GasAs 660nm 4 J/cm².
  Arms: Comparador ativo: LG1 + curativo
Device: LG2 — Application of LASER GasAs 660nm 8 J/cm².
  Arms: Comparador ativo: LG2 + curativo
Device: LG3 — Application of LASER GasAs 660nm 12 J/cm².
  Arms: Comparador ativo: LG3 + curativo
Procedure: Dressing — Application of Helianthus annuus oil dressing.

SUMMARY:
Diabetes mellitus consists of a heterogeneous group of metabolic disorders that have hyperglycemia in common, resulting from defects in insulin action, insulin secretion, or both. Diabetes mellitus has gained increasing importance and is considered one of the main themes of global health problems due to the damage caused to quality of life, public health and the epidemiological picture presented. Among the complications are diabetic foot ulcers, with higher prevalence in the lower limbs, they are classified as loss of skin continuity, which can reach from the epidermis to deep structures such as muscles, bones and tendons.

DETAILED DESCRIPTION:
100 volunteers will be recruited and the research will be carried out through the Integrated Center of Medical Specialties (CIEM) - Polyclinic, through referral from the specialist in vascular surgery after a thorough examination of the feet. Volunteers of both sexes, aged over 18 years, DM and diabetic ulcers will be admitted. Volunteers who present any autoimmune disease, concomitant psychiatric disorders or contraindications to the treatment methods adopted by the research will be excluded. Inclusion in the study will take place after signing the informed consent forms, after approval by the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patients with diabetic foot ulcers;
* Patients aged 18 and over.

Exclusion Criteria:

* Patients with autoimmune diseases
* Patients with concomitant psychiatric disorders
* Patients with contraindications to treatment methods
* Patients with infected diabetic foot ulcers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in the ulcer area | Before intervention starts, 5th and 10th week of intervention.
  Measure of ulcer area change.
Change in complete ulcer healing | Before intervention starts, 5th and 10th week of intervention.
  Change in the percentage of complete ulcer healing.

CONTACTS AND LOCATIONS:
Overall Officials: Vinicius Saura Cardoso, Principal Investigator — Federal University of Piaui
Locations (1):
- Federal University of Piaui, Parnaíba, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bezerra Miranda M, Silva Barros AC, Veloso Coelho L, Barbosa da Rocha R, Antonio Kato da Silva B, Ahmad Hazime F, Tanuri Magalhaes A, Saura Cardoso V. Dose-response and efficacy of 660-nanometer low-level laser therapy in healing diabetic foot ulcers: a randomized, double-blind, clinical trial. Lasers Med Sci. 2025 Oct 1;40(1):399. doi: 10.1007/s10103-025-04641-2. PMID 41028567